CLINICAL TRIAL: NCT00518310
Title: Azathioprine and Prednisone in the Treatment of Idiopathic Pulmonary Fibrosis: a Randomized, Double-Blind, Controlled Study
Brief Title: Azathioprine and Prednisone in the Treatment of Idiopathic Pulmonary Fibrosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Thorax National Institute (Other Government)
Collaborators: Sociedad Chilena de Enfermedades Respiratorias (Unknown); Servicio de Salud Metropolitano Oriente, Ministerio de Salud de Chile (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10351
Record Dates: First submitted 2007-08-16; First posted 2007-08-20 (Estimated); Last update posted 2007-08-20 (Estimated); Status verified 2007-08

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Interstitial lung disease; Idiopathic pulmonary fibrosis; Usual interstitial pneumonia; Cryptogenic fibrosing alveolitis; Therapy; Azathioprine; Steroids; Glucocorticoids; Corticosteroids; Prednisone
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Lung Diseases, Interstitial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 0 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- 1 (Active Comparator): Azathiprine Prednisone
  Interventions: Drug: AZAPRED

INTERVENTIONS:
Drug: Placebo
  Arms: 0
Drug: AZAPRED — The initial dose of prednisone will be 0.5 mg/kg/day for 4 weeks, then 0.25 mg/kg/day for 8 weeks. The dose will continue to decrease at a rate of 5 to 10 mg per week, to a dose of 0.25 or 0.125 mg/kg/day. Azathioprine will be given at a dose of 2-3 mg/kg/day (max 100 mg).
  Arms: 1

SUMMARY:
Idiopathic pulmonary fibrosis (IPF) is a diffuse lung disease, associated with the histological appearance of usual interstitial pneumonia (UIP), with an inexorably deteriorating clinical course. Prognosis is poor, reported median survival is less than 3 years. The prevalence is estimated as being 3 to 10 per 100.000 in different Western populations. To date, no pharmacological therapy has been proven to alter or reverse the pathogenic process of IPF. Most treatments trials have been observational case series of small patient populations and very few have been randomized, prospective and placebo-controlled.

Two recent Cochrane reviews investigated the role of corticosteroids and other immunomodulatory agents and concluded that there is no evidence for their use in IPF. Most current therapies are targeted to suppress the inflammatory component of the disease, based on the theory that it would be chronic alveolar inflammation which leads to parenchymal remodeling and fibrosis. Recently, a hypothesis that has gained acceptance suggests that fibrosis may result directly from alveolar injury, promoting an abnormal fibrogenic repair mediated by fibroblasts and myofibroblasts.

One of the cytotoxic agents most widely used and better tolerated in the management of IPF is azathioprine. Based upon limited data available and from a single small high quality randomized controlled trial (RCT), this drug appears to confer, given in conjunction with prednisone, a marginal long term survival advantage. Since this combination therapy is associated serious adverse effect, we planned to design a trial of low dose corticosteroid and azathioprine versus placebo in management of IPF, evaluating progression-free survival.

Our study hypothesis is: Combined therapy with azathioprine and corticosteroids improves progression-free survival in patients with the diagnosis of IPF.

DETAILED DESCRIPTION:
We will evaluate all adult patients consecutively referred from March 2005 to the Instituto Nacional del Tórax (Thorax National Institute), Santiago, Chile for diagnostic evaluation of Pulmonary Fibrosis. The routine evaluation will include, when indicated, the following steps:

* History:
* Age
* Genre
* Duration of symptoms before first consultation
* Smoking status
* Search for collagen vascular disease
* Family history of pulmonary fibrosis
* Occupational exposures
* Drug ot toxic exposures
* Physical examination: search of crackles and finger clubbing.
* Laboratory data:
* Complete blood bell count
* BUN
* Creatinine
* Liver enzymes
* Antinuclear antigens
* Erythrocyte sedimentation rate
* Rheumatoid factor
* HIV
* Antineutrophil cytoplasmic antibody (in appropiate clinical setting)
* Antiglomerular basement antibody (in appropiate clinical setting)
* Modified Medical Research Council Dyspnea Scale (MMRC) (10)
* Chronic Respiratory Questionnaire (CRQ) (11)
* Pulmonary function tests:
* Spirometry
* Plethismographic lung volumes
* DLco
* Composite physiologic index (12)
* Exercise testing:
* Six-Minute Walk Test (6MWT)
* Resting and 6 minute SpO2
* Presence or absence of desaturation to 88% or lower at the end of the six minute walk (13)
* Walked distance
* Pre and post modified Borg dyspnea scores
* Timed walk test (14)
* Arterial blood gas analysis in rest and exercise, calculating the difference between alveolar and arterial oxygen tension (P(A-a)O2) at rest and after exercise.
* Radiologic studies:
* Chest radiography
* HRCT:
* Definite or probable idiopathic pulmonary fibrosis (15):

  * Definitive criteria: presence of lung volume reduction, reticular abnormalities, traction bronchiectasis, or both, with a basal and peripheral predominance; the presence of honeycombing with a basal and peripheral predominance; and the absence of atypical features of usual interstitial pneumonia - micronodules, peribronchovascular nodules, consolidation, isolated (nonhoneycombing) cysts, ground-glass attenuation (or if present, less extensive than the reticular opacity), and mediastinal adenopathies (or if present, too limited to be visible on a chest radiography).
  * Probable criteria: presence of a bilateral, predominantly basal and subpleural reticular pattern with subpleural cysts (honeycombing), traction bronchiectasis, or both in the absence of atypical features of UIP.
* Scoring of the extent of lung fibrosis (16).
* Bronchoscopy:
* Bronchoalveolar lavage: cellular analysis and CD4/CD8 ratio.
* Transbronchial biopsy.
* Surgical lung biopsy:
* Number
* Site/Side
* Type of surgery: open vs thoracoscopic
* Histologic features (3)

Those patients with IPF diagnosed on the basis of clinical and radiographic criteria alone according to the ATS/ERS consensus committee (3), and/or with a biopsy proven histological pattern of UIP, will be selected to the randomization process, after they have signed the written informed consent.

ELIGIBILITY:
Inclusion Criteria:

* 45 and 79 years of age.
* Clinical symptoms of IPF for at least 3 months.
* Forced vital capacity (FVC) between 50 to 90% of the predicted value.
* DLco at least 35% of the predicted value.
* PaO2 > 55 mm Hg while breathing ambient air at rest.
* High-resolution computed tomography (HRCT) showing definite or probable criteria of IPF.

Exclusion Criteria:

* Clinically significant exposure to known fibrogenic agents (birds, molds, hot tubes, asbestos, radiation and drugs known to cause pulmonary fibrosis (amiodarone, nitrofurantoin, bleomicin,etc)).
* History of neurofibromatosis, Hermansky-Pudlak syndrome, metabolic storage disorders, etc.
* History of fever, weight loss, myalgias, arthralgias, skin rash, arthritis.
* Active infection within one week before enrollment.
* Alternative cause of interstitial lung disease.
* Ratio of the forced expiratory volume in one second (VEF1) to FVC of less than 0.6 after the use of a bronchodilator.
* Residual volume more than 120% of the predicted value (when available).
* More than 20% of lymphocytes or eosinophils in bronchoalveolar lavage (BAL) (when available).
* Granulomas, infection or malignancy in the transbronchial or surgical biopsy (when available).
* Previous therapy with azathioprine, prednisolone (>0.5 mg/kg/day or more for at least 3 months), cyclophosphamide or novel biotech drugs.
* Unstable cardiovascular or neurologic disease.
* Uncontrolled diabetes.
* Pregnancy.
* Lactation.
* Likelihood of death, as predicted by the investigator, within the next year.
* White cell blood count < 4000/mm3.
* Platelet count < 100000/mm3.
* Hematocrit < 30% or > 59%.
* Liver enzymes more than 3 times the upper limit of the normal range.
* Creatinine level > 1.5 mg/dL.
* Albumin level < 3 g/dL.
* Refusal to sign informed consent by patient or guardian.

Ages: 45 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-05; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival, defined as free of death or a decrease from baseline in the FVC of at least 10%. | 2 years

SECONDARY OUTCOMES:
Number of Acute Exacerbations of IPF. | 2 years
Health Related Quality of life, measured with the Chronic Questionnaire (CRQ). | 2 years
PO2 at rest and at exercise from baseline. | 2 years
P(A-a)O2 at rest and at exercise from baseline. | 2 years
Predicted FEV1 from baseline. | 2 years
Forced expiratory volume in one second (FEV1) to FVC from baseline. | 2 years
Plethysmographic lung volumes from baseline. | 2 years
Diffusion capacity for carbon monoxide (DLco) from baseline. | 2 years
Six-Minute Walk test, from baseline: resting and 6 minute SpO2, presence or absence of desaturation to 88% or lower at the end of the six minute walk, walked distance d. Pre and post modified Borg dyspnea scores | 2 years
Scoring of extent of lung fibrosis on HRCT, according to two independent chest radiologists, form baseline. | 2 years
Number and severity of adverse effects. | 2 years
Number of protocol drop outs. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Florenzano Matías, MD, Principal Investigator — Clínica Las Condes
Locations (1):
- Instituto Nacional del Tórax, Santiago, RM, Chile